



## INFORMED CONSENT FOR THE STUDY

| Title of the study: "Implementation in Colorectal Surgery of a new modular and open robotic platform. Pilot project." Protocol code: COLOROBOT-ELX24 Principal investigator: | |
|---|---|
| D. /D <sup>a</sup> : | with DNI: |
| <ul> <li>which I am invited to participate.</li> <li>That I know and assume the risks and/or consection.</li> <li>That I have read and understood this writing asked all the questions I thought appropriate an I accept that my personal data will be used to past I understand that my participation is voluntary.</li> <li>I have received a signed copy of this informed consecutive.</li> </ul> | I am satisfied with the information received, I have ad all my doubts have been clarified. articipate in the study for research purposes. |
| Signature of the physician/investigator | Signature of the patient |
| Dr./a: | D. /D <sup>a</sup> : |
| D. /Da: | , with DNI: give my consent to have the |
| Revocation of consent: D. /Da: I REVOCATE the consent previously given to carry out this pro | , con DNI:ocedure of my own free will. |
| Signature of the patient Date: | Signature of the physician/investigator Date: |
| Signature of representative Date: | |